CLINICAL TRIAL: NCT01784068
Title: A Single-arm, Multicenter, Nilotinib Treatment-free Remission Study in Patients With BCR-ABL1 Positive Chronic Myelogenous Leukemia in Chronic Phase Who Have Achieved Durable Minimal Residual Disease (MRD) Status on First Line Nilotinib Treatment.
Brief Title: Nilotinib Treatment-free Remission Study in CML (Chronic Myeloid Leukemia) Patients
Acronym: ENESTfreedom
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CAMN107I2201; 2012-004092-40 (EudraCT Number)
Record Dates: First submitted 2013-01-30; First posted 2013-02-05 (Estimated); Results first posted 2021-01-14 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Chronic Myelogenous Leukemia
Keywords: AMN107; Ph+ CML-CP; chronic phase; nilotinib treatment; 2 years treatment; MR 4.5; Loss of MR 4; Loss of MMR; CML
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — nilotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Nilotinib followed by treatment-free (Experimental): Patients who received a minimum of 2 years of first line nilotinib treatment and with pre-screen PCR results in ≥ MR4.5 entered the consolidation phase of the study (52 weeks - nilotinib 300 mg BID). Patients with Minimal Residual Disease (MRD) at the end of this phase entered the Treatment-Free Remission (TFR) phase where no treatment was given. Non eligible patients will enter the continuation phase of the study. Patients with MRD at the end of the continuation phase will enter the TFR-2 phase of the study where no treatment is given. Non eligible patients will enter the prolonged continuation phase of the study. If at any time during TFR or TFR-2 the patient loses MMR, nilotinib treatment will be immediately re-initiated (nilotinib 300 mg BID).
  Interventions: Drug: Nilotinib followed by treatment-free

INTERVENTIONS:
Drug: Nilotinib followed by treatment-free — Nilotinib is being used as commercial available capsules (except in Japan where clinical supplies is used) of 150 mg and 200 mg strength. Treatment occurs during consolidation, continuation, prolonged continuation, re-initiation and re-initiation-2 phases of the study.
  Other Names: AMN107

SUMMARY:
The main purpose of the study was to investigate whether nilotinib treatment can be safely suspended with no recurrence of CML in selected patients who responded optimally on this treatment

DETAILED DESCRIPTION:
The Primary objective of this study was to determine the percentage of patients who were in MMR at 48 weeks after starting the TFR phase (patients who required re-initiation of treatment were considered as non-responders).

Nilotinib treatment consolidation phase (NTCS): Patients who satisfied all inclusion/exclusion criteria were enrolled in the consolidation phase and continued to receive nilotinib for 52 weeks. All patients were treated with the planned nilotinib dose 300 mg BID (or at a reduced dose level of 400 mg QD if required from the perspective of toxicity). In order for patients to be eligible for the TFR phase, they had to fulfill the protocol specific definition of durable MRD. The four last quarterly performed PCR assessments must have fulfilled the following criteria:

* The last assessment was MR4.5 (BCR-ABL ≤ 0.0032% IS)
* No assessment worse than MR4.0 (BCR-ABL >0.01% IS) and
* No more than two assessments between MR4.0 and MR4.5 (0.0032% IS<BCR-ABL ≤ 0.01% IS)

Nilotinib TFR phase: Patients who were eligible to enter in the TFR phase after completing the 52 weeks consolidation phase, stopped taking nilotinib on the first day of the TFR phase. Duration of this phase was up to 10 years after the last patient enters in the TFR phase. BCR-ABL levels were monitored every four weeks during the first 48 weeks, every six weeks for the following 48 weeks and every 12 weeks during the last period.

Nilotinib treatment re-initiation (NTRI) phase: If a patient had a loss of MMR (BCR-ABL >0.1% IS) in the TFR phase, the patient restarted nilotinib treatment. Patients were on nilotinib treatment for up to 10 years after the last patient entered the nilotinib TFR phase. Patients who required re-initiation of nilotinib treatment were monitored for the BCR-ABL level every four weeks for the first 24 weeks and then every 12 weeks thereafter in patients who regained MMR. The frequency of BCR-ABL monitoring in patients not regaining MMR within the first 24 weeks after re-initiation of treatment was at least every 12 weeks or more frequently as clinically indicated.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients ≥ 18 years of age
* Minimum of 2 calendar years of nilotinib treatment with at least the last 12 months of nilotinib treatment prior to pre-screening at approved total daily dose of 600 mg BID or at a reduced dose of 400 mg QD if required from the perspective of tolerance for BCR-ABL positive CML in documented chronic phase at the time of diagnosis
* Evidence of typical BCR-ABL transcripts (b3a2 and/or b2a2) at the time of CML-CP diagnosis i.e. prior to first start of TKI treatment which are amenable to standardized RT-PCR quantification"
* Patient in MR4.5 at prescreening at Novartis designated lab
* ECOG performance status of 0-2
* Adequate end organ function as defined by:

  * Direct bilirubin ≤ 1.5 x ULN except for i) patients with documented Gilbert's syndrome for whom any bilirubin value is allowed and ii) for patients with asymptomatic hyperbilirubinemia (liver transaminases and alkaline phosphatase within normal range).
  * SGOT(AST) and SGPT(ALT) ≤ 3 x ULN i.e. equivalent to ≤ Grade 1 NCI-CTCAE v.4.03
  * Serum lipase ≤ 2 x ULN i.e. equivalent to ≤ Grade 2 NCI-CTCAE v.4.03
  * Alkaline phosphatase ≤ 2.5 x ULN
  * Serum creatinine < 1.5 x ULN
* Patients must have the following electrolyte values within normal limits or corrected to be within normal limits with supplements prior to first dose of study medication:

  * Potassium (suggested keep to prevent issues with QT and/or rhythm abnormalities)
  * Magnesium (suggested keep to prevent issues with QT and/or rhythm abnormalities)
  * Total calcium (corrected for serum albumin)
* Patients must have normal marrow function as defined:

  * Absolute Neutrophil Count (ANC) ≥ 1.5 x 10E9/L
  * Hemoglobin ≥ 9.0 g/dL
  * Platelets ≥ 100 x 10E9/L
* Documented chronic phase CML must meet all the criteria defined by:

  * < 15% blasts in peripheral blood and bone marrow,
  * < 30% blasts plus promyelocytes in peripheral blood and bone marrow,
  * < 20% basophils in the peripheral blood,
  * ≥ 100 x 109/L (≥ 100,000/mm3) platelets,
  * No evidence of extramedullary leukemic involvement, with the exception of hepatosplenomegaly
* Patients must tolerate a minimum total daily dose of nilotinib of 400 mg

Exclusion Criteria:

* Previous treatment with BCR-ABL inhibitors other than nilotinib for more than a total cumulative duration of 4 weeks
* Previous treatment with alpha-interferon of any duration
* Previous anticancer agents for CML other than nilotinib except for cytoreduction after CML diagnosis until up to 4 weeks after first dose of nilotinib
* Known second chronic phase of CML after previous progression to AP/BC
* Poorly controlled diabetes mellitus (defined as HbA1c > 9%)
* Impaired cardiac function including any one of the following:

  * LVEF < 45% or below the institutional lower limit of the normal range (whichever is higher)
  * Inability to determine the QT interval on ECG, except for patients with evidence of measurable QT interval at the time of CML diagnosis (e.g. prior to first start of TKI treatment) and who have no documented clinical signs of cardiovascular disease and/or clinical signs of conduction abnormality.
  * Complete left bundle branch block
  * Right bundle branch block plus left anterior or posterior hemiblock
  * Use of a ventricular-paced pacemaker
  * Congenital long QT syndrome or a known family history of long QT syndrome
  * History of or presence of clinically significant ventricular or atrial tachyarrhythmias
  * Clinically significant resting bradycardia
  * QTc > 450 msec on the average of three serial baseline ECG (using the QTcF formula). If QTcF > 450 msec and electrolytes are not within normal ranges, electrolytes should be corrected and then the patient re-tested for QTc.This exclusion criterion is not applicable for patients with non-measurable QT interval who have evidence of measurable QT interval at the time of CML diagnosis (e.g. prior to first start of TKI treatment) and who have no documented clinical signs of cardiovascular disease and/or clinical signs of conduction abnormality.
  * History or clinical signs of myocardial infarction within 1 year of study entry
  * History of unstable angina within 1 year of study entry
  * Other clinically significant heart disease (e.g. congestive heart failure, cardiomyopathy or uncontrolled hypertension)
* History of acute pancreatitis within 1 year of study entry or past medical history of chronic pancreatitis
* Known presence of significant congenital or acquired bleeding disorder unrelated to cancer
* Severe and/or uncontrolled concurrent medical disease that in the opinion of the investigator could cause unacceptable safety risks or compromise compliance with the protocol (e.g. uncontrolled diabetes, uncontrolled infection)
* History of another active malignancy within 5 years prior to study entry with the exception of previous or concomitant basal cell skin cancer and previous carcinoma in situ treated curatively
* Treatment with other investigational agents (defined as not used in accordance with the approved indication) within 4 weeks of Day 1
* Patients who have not recovered from prior surgery
* Patients actively receiving therapy with strong CYP3A4 inhibitors and/or inducers, and the treatment cannot be either discontinued or switched to a different medication prior to starting study drug.
* Patients actively receiving therapy with herbal medicines that are strong CYP3A4 inhibitors and/or inducers, and the treatment cannot be either discontinued or switched to a different medication prior to starting study drug. These herbal medicines may include Echinacea, (including E. purpurea, E. angustifolia and E. pallida), Piperine, Artemisinin, St. John's Wort, and Ginkgo.
* Patients who are currently receiving treatment with any medications that have the potential to prolong the QT interval and the treatment cannot be either safely discontinued or switched to a different medication prior to starting study drug. (see http://www.torsades.org/medical-pros/drug-lists/printable-drug-list.cfm for a list of agents that prolong the QT interval)
* Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of study drug (e.g. ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, small bowel resection, or gastric bypass surgery)
* Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test.
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception during the study and for 14 days after the final dose of nilotinib. Highly effective contraception is defined as either:

  * Total abstinence (when this is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception
  * Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy) or tubal ligation at least six weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment.
  * Male sterilization (at least 6 months prior to enrolling). For female patients on the study the vasectomized male partner should be the sole partner for that patient.
  * Use of a combination of any two of the following:

    1. Use of oral, injected or implanted hormonal methods of contraception or other forms of hormonal contraception that have comparable efficacy (failure rate <1%), for example hormone vaginal ring or transdermal hormone contraception.
    2. Placement of an intrauterine device (IUD) or intrauterine system (IUS)
    3. Barrier methods of contraception: Condom or Occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/vaginal suppository.

In case of use of oral contraception women should have been stable on the same pill for a minimum of 3 months before taking study treatment Women are considered post-menopausal and not of child bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks prior to enrolling. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of child bearing potential.

If a study patient becomes pregnant or suspects being pregnant during the study or within 30 days after the final dose of nilotinib, the Study Doctor needs to be informed immediately and ongoing study treatment with nilotinib has to be stopped immediately.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 215 (Actual)
Dates: Start 2013-03-19 (Actual); Primary Completion 2016-05-31 (Actual); Study Completion 2025-01-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (104):
- United States (10):
  - Florida Cancer Specialists, Fort Myers, Florida
  - Lakes Research, Miami Lakes, Florida
  - H Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Cancer Center of Kansas, Wichita, Kansas
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan Kettering, New York, New York
  - Oregon Health Sciences University, Portland, Oregon
  - Cancer Centers of the Carolinas, Greenville, South Carolina
  - Tennessee Oncology PLLC, Chattanooga, Tennessee
  - Community Cancer Trials of Utah, Ogden, Utah
- Novartis Investigative Site, Buenos Aires, Argentina
- Austria (4):
  - Novartis Investigative Site, Graz
  - Novartis Investigative Site, Rankweil
  - Novartis Investigative Site, Salzburg
  - Novartis Investigative Site, Vienna
- Belgium (6):
  - Novartis Investigative Site, Sint-Niklaas, Oost Vlaanderen
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Charleroi
  - Novartis Investigative Site, Ghent
  - Novartis Investigative Site, Kortrijk
  - Novartis Investigative Site, Liège
- Novartis Investigative Site, Varna, Bulgaria
- Colombia (2):
  - Novartis Investigative Site, Bogota, Cundinamarca
  - Novartis Investigative Site, Montería
- Novartis Investigative Site, Aarhus N, Denmark
- France (11):
  - Novartis Investigative Site, Bayonne, Bayonne Cedex
  - Novartis Investigative Site, Saint Priest En Jarez, Pays de la Loire Region
  - Novartis Investigative Site, Bordeaux
  - Novartis Investigative Site, Brest
  - Novartis Investigative Site, Corbeil-Essonnes
  - Novartis Investigative Site, Dunkirk
  - Novartis Investigative Site, Grenoble
  - Novartis Investigative Site, Nantes
  - Novartis Investigative Site, Rouen
  - Novartis Investigative Site, Strasbourg
  - Novartis Investigative Site, Toulouse
- Germany (20):
  - Novartis Investigative Site, Freiburg im Breisgau, Baden-Wurttemberg
  - Novartis Investigative Site, Mannheim, Baden-Wurttemberg
  - Novartis Investigative Site, Frankfurt am Main, Hesse
  - Novartis Investigative Site, Düsseldorf, North Rhine-Westphalia
  - Novartis Investigative Site, Leipzig, Saxony
  - Novartis Investigative Site, Lübeck, Schleswig-Holstein
  - Novartis Investigative Site, Jena, Thuringia
  - Novartis Investigative Site, Aachen
  - Novartis Investigative Site, Bayreuth
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bonn
  - Novartis Investigative Site, Bottrop
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Düsseldorf
  - Novartis Investigative Site, Goslar
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Magdeburg
  - Novartis Investigative Site, Mainz
  - Novartis Investigative Site, Stuttgart
  - Novartis Investigative Site, Ulm
- Novartis Investigative Site, Athens, Greece
- Hungary (2):
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Szeged
- Ireland (2):
  - Novartis Investigative Site, Dublin
  - Novartis Investigative Site, Galway
- Italy (13):
  - Novartis Investigative Site, Ancona, AN
  - Novartis Investigative Site, Brescia, BS
  - Novartis Investigative Site, Cona, FE
  - Novartis Investigative Site, Florence, FI
  - Novartis Investigative Site, Genova, GE
  - Novartis Investigative Site, Nuoro, NU
  - Novartis Investigative Site, Perugia, PG
  - Novartis Investigative Site, Reggio Calabria, RC
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Orbassano, TO
  - Novartis Investigative Site, Terni, TR
  - Novartis Investigative Site, Napoli
  - Novartis Investigative Site, Novara
- Japan (12):
  - Novartis Investigative Site, Kashiwa, Chiba
  - Novartis Investigative Site, Sapporo, Hokkaido
  - Novartis Investigative Site, Sagamihara, Kanagawa
  - Novartis Investigative Site, Ōsaka-sayama, Osaka
  - Novartis Investigative Site, Suita, Osaka
  - Novartis Investigative Site, Saga, Saga-ken
  - Novartis Investigative Site, Kawagoe, Saitama
  - Novartis Investigative Site, Shimotsuga Gun, Tochigi
  - Novartis Investigative Site, Bunkyo-ku, Tokyo
  - Novartis Investigative Site, Shinjuku Ku, Tokyo
  - Novartis Investigative Site, Akita
  - Novartis Investigative Site, Kumamoto
- Novartis Investigative Site, Groningen, Netherlands
- Poland (2):
  - Novartis Investigative Site, Gdansk
  - Novartis Investigative Site, Warsaw
- Spain (10):
  - Novartis Investigative Site, Terrassa, Catalonia
  - Novartis Investigative Site, Ourense, Galicia
  - Novartis Investigative Site, Pamplona, Navarre
  - Novartis Investigative Site, Oviedo, Principality of Asturias
  - Novartis Investigative Site, San Cristóbal de La Laguna, Santa Cruz De Tenerife
  - Novartis Investigative Site, Barakaldo, Vizcaya
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Las Palmas de Gran Canaria
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Tarragona
- Sweden (3):
  - Novartis Investigative Site, Lund
  - Novartis Investigative Site, Stockholm
  - Novartis Investigative Site, Uppsala
- United Kingdom (2):
  - Novartis Investigative Site, Cardiff
  - Novartis Investigative Site, Oxford

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 215 patients were actually enrolled in the NTCS (nilotinib treatment consolidation) phase. 190 of the 215 patients completed 52 weeks of nilotinib treatment in the NTCS phase and entered the treatment-free remission (TFR) phase.
Pre-assignment Details: Approximately 175 patients were planned to be enrolled into the study.
Groups:
- NTCS Phase: Patients who received a minimum of two years of first line nilotinib treatment and with BCR-ABL1 transcript level of MR4.5 entered consolidation phase of the study (52 weeks of nilotinib 300 mg BID)
- TFR Phase: Patients with Minimal Residual Disease (MRD) at the end of consolidation phase entered the Treatment-Free Remission (TFR) phase where no treatment was given
Period: NTCS Phase
Arm/Group | NTCS Phase | TFR Phase
Started | 215 | 0
NTRI Phase | 86 | 0
NTCT Phase | 13 | 0
TFR-2 Phase | 8 | 0
NTCT-P Phase | 2 | 0
NTRI-2 | 0 | 0
Completed (Completed = Still on Study Phase which means a patient has no end of study phase completion CRF page as of data Cut-off date: 30-NOV-2015) | 0 | 0
Not Completed | 215 | 0
Not completed — Adverse Event | 5 | 0
Not completed — Physician Decision | 2 | 0
Not completed — Patient/guardian decision | 3 | 0
Not completed — Death | 2 | 0
Not completed — Completed phase = discontinuation of study except for TFR and TFR2 phases | 203 | 0
Period: TFR Phase
Arm/Group | NTCS Phase | TFR Phase
Started | 0 | 190
Completed | 0 | 97
Not Completed | 0 | 93
Not completed — Physician Decision | 0 | 1
Not completed — Patient/guardian decision | 0 | 3
Not completed — Death | 0 | 1
Not completed — Lack of Efficacy | 0 | 88

BASELINE CHARACTERISTICS:
Population: Safety Set: Safety set included all patients who received at least one dose of study medication.
Arm/Group | NTCS Phase
Number analyzed (Participants) | 215
Age, Continuous [Median (Full Range); unit: years] | 54.0 [21 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 102
  Male | 113
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 189
  Asian | 20
  Unknown | 3
  Native American | 1
  Other | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Who Are in MMR (Major Molecular Response) at 48 Weeks After Starting the Treatment-free Remission (TFR) Phase
Description: Primary endpoint was the percentage of participants who were in MMR at 48 weeks after starting the TFR phase and is calculated by dividing the number of patients with MMR at 48 weeks after starting the TFR phase with no loss of MMR and no re-initiation of nilotinib therapy in the first 48 weeks after starting the TFR phase by the number of patients who entered the TFR phase. Patients who required re-initiation of treatment were considered as non-responders.
Time Frame: 48 weeks
Population: FAS: The FAS included the 190 patients who completed 52 weeks of nilotinib treatment in the NTCS phase and entered TFR phase
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | TFR Phase
Number analyzed (Participants) | 190
Percentage of participants | 51.6 [44.2 to 58.9]

2. Secondary Outcome: Percentage of Patients Who Are in MR4.5 (BCR-ABL ≤ 0.0032% IS) at 48 Weeks After Starting the TFR Phase
Description: Proportion of patients who are in MR4.5 at 48 weeks after starting the TFR phase is calculated by dividing the number of patients with MR4.5 at 48 weeks after starting the TFR phase with no loss of MR4.5 and no re-initiation of nilotinib therapy in the first 48 weeks after starting the TFR phase by the number of patients who entered the TFR phase. Patients who required re-initiation of treatment will be considered as non-responders. MR4.5 = log reductions of the BCR-ABR transcript load in blood as a measurement of deep molecular response of the CML clone to treatment.
Time Frame: 48 weeks
Reporting Status: Not Posted, anticipated posting 2026-01

3. Secondary Outcome: Percentage of Patients Who Are in MMR at 96, 144,192, 264 Weeks and at the End of 6, 7, 8, 9 and 10 Years After Starting the TFR Phase
Description: Proportion of patients who are in MMR at 96, 144, 192, 264 weeks and at the end of 6, 7, 8, 9 and 10 years after starting the TFR phase is calculated by dividing the number of patients with MMR at 96, 144, 192, 264 weeks and at the end of 6, 7, 8, 9 and 10 years after starting the TFR phase with no loss of MMR and no re-initiation of nilotinib therapy in the first 96, 144, 192, 264 weeks and at the end of 6, 7, 8, 9 and 10 years after starting the TFR phase by the number of patients who entered the TFR phase. Patients who required re-initiation of treatment will be considered as non-responders
Time Frame: 96, 144, 192, 264 weeks, end of 6, 7, 8, 9 and 10 years
Reporting Status: Not Posted, anticipated posting 2026-01

4. Secondary Outcome: Percentage of Patients Who Are in MR4.5 at 96, 144, 192, 264 Weeks and at the End of 6, 7, 8, 9 and 10 Years After Starting the TFR Phase
Description: Proportion of patients who are in MR4.5 at 96, 144, 192, 264 weeks and at the end of 6, 7, 8, 9 and 10 years after starting the TFR phase is calculated by dividing the number of patients with MR4.5 at 96, 144, 192, 264 weeks and at the end of 6, 7, 8, 9 and 10 years after starting the TFR phase with no loss of MR4.5 and no re-initiation of nilotinib therapy in the first 96, 144, 192, 264 weeks and at the end of 6, 7, 8, 9 and 10 years after starting the TFR phase by the number of patients who entered the TFR phase. Patients who required re-initiation of treatment will be considered as non-responders
Time Frame: 96, 144, 192, 264 weeks, end of 6, 7, 8, 9 and 10 years
Reporting Status: Not Posted, anticipated posting 2026-01

5. Secondary Outcome: Percentage of Patients in MMR at 48, 96, 144, 192, 264 Weeks and at the End of 6, 7, 8, 9 and 10 Years After Starting the TFR Phase of Nilotinib
Description: Proportion of patients who are in MMR at 48, 96, 144, 192, 264 weeks and at the end of 6, 7, 8, 9 and 10 years after starting the TFR phase is calculated by dividing the number of patients with MMR at 48, 96, 144, 192, 264 weeks and at the end of 6, 7, 8, 9 and 10 years after starting the TFR phase by the number of patients who entered the TFR phase. Patients who are re-initiated with nilotinib but have less than 12 weeks of re-initiation of treatment will be excluded from the analysis
Time Frame: 48, 96, 144, 192, 264 weeks and at the end of 6, 7, 8, 9 and 10 years
Reporting Status: Not Posted, anticipated posting 2026-01

6. Secondary Outcome: Percentage of Patients in MR4.5 at 48, 96, 144, 192, 264 Weeks and at the End of 6, 7, 8, 9 and 10 Years After Starting the TFR Phase of Nilotinib
Description: Proportion of patients who are in MR4.5 at 48, 96, 144, 192, 264 weeks and at the end of 6, 7, 8, 9 and 10 years after starting the TFR phase is calculated by dividing the number of patients with MR4.5 at 48, 96, 144, 192, 264 weeks and at the end of 6, 7, 8, 9 and 10 years after starting the TFR phase by the number of patients who entered the TFR phase. Patients who are re-initiated with nilotinib but have less than 12 weeks of re-initiation of treatment will be excluded from the analysis
Time Frame: 48, 96, 144, 192, 264 weeks, end of 6, 7, 8, 9 and 10 years
Reporting Status: Not Posted, anticipated posting 2026-01

7. Secondary Outcome: Percentage of Patients Who Achieve MMR Within 12 Weeks of Re-treatment With Nilotinib
Description: Proportion of patients who achieve MMR within 12 weeks of re-initiation of nilotinib is calculated by dividing the number of patients who are in MMR at least at one assessment within 12 weeks after re-start of nilotinib treatment by the number of patients who are re-initiated for at least 12 weeks
Time Frame: 12 weeks
Reporting Status: Not Posted, anticipated posting 2026-01

8. Secondary Outcome: Kinetics of BCR-ABL Transcript After Re-start of Nilotinib Therapy
Description: Descriptive statistics of BCR-ABL levels (IS) over time after re-start of nilotinib therapy up to 528 weks after the last patient has entered TFR
Time Frame: Every 4 weeks up to week 24 and every 12 weeks thereafter up to 528 weeks after last patient has entered the TFR
Reporting Status: Not Posted, anticipated posting 2026-01

9. Secondary Outcome: Duration of Re-initiated Treatment Required to Regain MMR After Loss of MMR
Description: Defined as time from date of start of re-initiation of treatment after loss of MMR to the date of first achievement of MMR. Patients who do not regain MMR after re-initiation of treatment on or before the cut-off date, duration will be censored at the date of last PCR assessment
Time Frame: Every 4 weeks up to week 24 and every 12 weeks thereafter up to 528 weeks after the last patient has entered TFR
Reporting Status: Not Posted, anticipated posting 2026-01

10. Secondary Outcome: Duration of Re-initiated Treatment Required to Regain MR4.5 After Loss of MMR
Description: Defined as the time from start of re-initiation of treatment after loss of MMR to the first achievement of MR4.5. Patients who do not regain MR4.5 after re-initiation of treatment on or before the cut-off date, duration will be censored at the date of last PCR assessment
Time Frame: Every 4 weeks up to week 24 and every 12 weeks thereafter up to 528 weeks after the last patient has entered TFR
Reporting Status: Not Posted, anticipated posting 2026-01

11. Secondary Outcome: Treatment-free Survival (TFS) After the Start of the TFR Phase
Description: TFS is defined as the time from the start of the TFR phase to the earliest occurrence of loss of MMR, re-initiation of treatment due to any cause, progression of AP/BC or death due to any cause. For patients without any event on or before the cut-off date, survival time will be censored at the date of their last assessment (PCR, cytogenetic, hematologic or extramedullary). A TFS sensitivity analysis will be conducted to consider discontinuation from TFR phase due to any reason as a TFS event, in addition to the TFS events as defined above.
Time Frame: Every 4 weeks in the first period of 48 weeks of the TFR, every 6 weeks in the second period of 48 weeks in TFR and every 12 weeks in the last period of 432 weeks of the TFR
Reporting Status: Not Posted, anticipated posting 2026-01

12. Secondary Outcome: Progression-free Survival (PFS) After the Start of the TFR Phase
Description: PFS is defined as the time from the start of the TFR phase to the earliest occurrence of progression to AP/BC or death due to any cause. For patients without any event on or before the cut-off date, survival time will be censored at the date of their last assessment (cytogenetic, hematologic or extramedullary) for patients who are still on study and at the date of last contact for patients who are in follow-up
Time Frame: Every 4 weeks in the first period of 48 weeks of the TFR, every 6 weeks in the second period of 48 weeks of TFR and every 12 weeks in the last period of 432 weeks of the TFR
Reporting Status: Not Posted, anticipated posting 2026-01

13. Secondary Outcome: Overall Survival (OS) After the Start of the TFR Phase
Description: OS is defined as the time from start of the TFR phase to death due to any cause. For patients without any event on or before the cut-off date, survival time will be censored at the date of their last assessment for patients who are still on study and at the date of last contact for patients who are in follow-up
Time Frame: as for outcome 12
Reporting Status: Not Posted, anticipated posting 2026-01

14. Secondary Outcome: Safety Profile During the Nilotinib Treatment Consolidation Phase, During the TFR Phase and During Re-initiation Treatment With Nilotinib
Description: Safety profile includes type, frequency and severity of adverse events, laboratory abnormalities and clinically notable ECG and other safety parameters during the nilotinib treatment consolidation phase, during the TFR phase and during re-initiation of treatment with nilotinib
Time Frame: Every 4 weeks in treatment consolidation and during the first 24 weeks of the re-initiation phase, every 12 weeks thereafter. Every 4, 6 and 12 weeks respectively in the first and second period of 48 weeks and in the last period of 432 weeks of the TFR
Reporting Status: Not Posted, anticipated posting 2026-01

15. Secondary Outcome: Proportion of Patients Who Develop T3151, E255K/V, Y253H, F359V/C/I Mutations on Study or Any Other BCR-ABL Mutations in Patients Who Lost MMR After Nilotinib Suspension
Description: Proportion will be calculated by dividing the number of patients who developT315I, E255K/V, Y253H, F359V/C/I mutations after nilotinib suspension by the number of patients who lost MMR
Time Frame: Every 3 months in patients who lost MMR until the result is negative or up to 528 weeks after the last patient entered TFR. On average 3 analyses (every 3 months or up to 264 weeks after the last patient has entered TFR.)
Reporting Status: Not Posted, anticipated posting 2026-01

16. Secondary Outcome: Percentage of Patients Who Are in Stable Response (MMR and MR4.5) After Achievement of That Response in Nilotinib Re-initiation Phase for 48, 96, 144, 192, 240, 288, 336, 384 and 432 Weeks, Based on Availability of Appropriate Data
Description: Proportion of patients who are in stable MMR/MR4.5 after achievement of that response in the nilotinib re-initiation phase for 48, 96, 144, 192, 240, 288, 336, 384 and 432 weeks, based on availability of appropriate data, is calculated by dividing the number of patients achieving MMR/MR4.5 any time during the nilotinib re-initiation phase and having the same response 48, 96, 144, 192, 240, 288, 336, 384 and 432 weeks after the first achievement of MMR/MR4.5, irrespective of whether there is loss of MMR in between, by the number of patients who achieved MMR/MR4.5 at any time during the nilotinib re-initiation phase
Time Frame: 48, 96, 144, 192, 240, 288, 336, 384 and 432 weeks
Reporting Status: Not Posted, anticipated posting 2026-01

ADVERSE EVENTS:
Time Frame: Adverse events were collected from first dose of study treatment until 30 days after the last dose of study treatment or the last day in the TFR/TFR-2 phase for approx. 26 months.
Description: Any sign or symptom that occurs during the study treatment plus 30 days post treatment.
Groups:
- NTRI Phase: If at any time during TFR phase the patient lost MMR, nilotinib treatment was to be immediately re-initiated (nilotinib 300 mg BID)
- NTCT Phase: Patients with no MRD at the end of consolidation phase entered the continuation phase of the study and continue with nilotinib 300 mg BID
- TFR-2 Phase: Patients with MRD at the end of the continuation phase entered the TFR-2 phase of the study where no treatment was given
- NTRI-2 Phase: If at any time during TFR phase or TFR-2 phase the patient lost MMR, nilotinib treatment was to be immediately re-initiated (nilotinib 300 mg BID)
- NTCT-P Phase: Patients with no MRD at the end of continuation phase entered the prolonged continuation phase of the study
- All Patients: All patients enrolled in the study
Arm/Group | NTCS Phase | TFR Phase | NTRI Phase | NTCT Phase | TFR-2 Phase | NTRI-2 Phase | NTCT-P Phase | All Patients
All-Cause Mortality (participants affected / at risk) | 2/215 | 1/190 | 2/86 | 0/13 | 0/8 | 0/0 | 0/2 | 5/215
Serious Adverse Events (participants affected / at risk) | 20/215 | 15/190 | 11/86 | 1/13 | 0/8 | 0/0 | 0/2 | 40/215
Other Adverse Events (participants affected / at risk) | 136/215 | 91/190 | 49/86 | 10/13 | 1/8 | 0/0 | 0/2 | 171/215
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NTCS Phase (N=215) | TFR Phase (N=190) | NTRI Phase (N=86) | NTCT Phase (N=13) | TFR-2 Phase (N=8) | NTRI-2 Phase (N=0) | NTCT-P Phase (N=2) | All Patients (N=215)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2
ANGINA PECTORIS (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
CARDIAC ARREST (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
CORONARY ARTERY DISEASE (Cardiac disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 2
MYOCARDIAL INFARCTION (Cardiac disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 2
IRIS NEOVASCULARISATION (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
ASCITES (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
GASTRIC ULCER (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
HAEMORRHOIDS (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
INGUINAL HERNIA (Gastrointestinal disorders) | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 3
NAUSEA (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
PANCREATITIS (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 2
CHEST PAIN (General disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2
DEATH (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
GENERALISED OEDEMA (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
CHOLELITHIASIS (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
HEPATOMEGALY (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
CONTRAST MEDIA ALLERGY (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
DRUG HYPERSENSITIVITY (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
DACRYOCYSTITIS (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
HERPES ZOSTER (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
PHARYNGEAL ABSCESS (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
TYPE 2 DIABETES MELLITUS (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
CHONDROPATHY (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 3
ROTATOR CUFF SYNDROME (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
BREAST CANCER IN SITU (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
MALIGNANT MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
MESOTHELIOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
RECTAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
THYROID NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
TRANSITIONAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
CEREBRAL INFARCTION (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
DIZZINESS (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
HEADACHE (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
MULTIPLE SCLEROSIS RELAPSE (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
SCIATICA (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
SYNCOPE (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
COMPLETED SUICIDE (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
HAEMORRHAGE URINARY TRACT (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
RENAL COLIC (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
URINARY INCONTINENCE (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
PERIPHERAL ARTERIAL OCCLUSIVE DISEASE (Vascular disorders) | 2 | 2 | 1 | 0 | 0 | 0 | 0 | 4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | NTCS Phase (N=215) | TFR Phase (N=190) | NTRI Phase (N=86) | NTCT Phase (N=13) | TFR-2 Phase (N=8) | NTRI-2 Phase (N=0) | NTCT-P Phase (N=2) | All Patients (N=215)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 9 | 6 | 3 | 0 | 0 | 0 | 0 | 15
DIARRHOEA (Gastrointestinal disorders) | 12 | 9 | 2 | 0 | 0 | 0 | 0 | 22
NAUSEA (Gastrointestinal disorders) | 7 | 2 | 3 | 1 | 0 | 0 | 0 | 10
VOMITING (Gastrointestinal disorders) | 6 | 5 | 1 | 0 | 0 | 0 | 0 | 11
FATIGUE (General disorders) | 9 | 6 | 4 | 0 | 0 | 0 | 0 | 18
INFLUENZA LIKE ILLNESS (General disorders) | 3 | 2 | 0 | 1 | 0 | 0 | 0 | 6
LOCALISED OEDEMA (General disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 2
GASTROENTERITIS (Infections and infestations) | 3 | 1 | 3 | 1 | 0 | 0 | 0 | 8
INFLUENZA (Infections and infestations) | 7 | 4 | 2 | 0 | 0 | 0 | 0 | 11
LARYNGITIS (Infections and infestations) | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 4
NASOPHARYNGITIS (Infections and infestations) | 22 | 17 | 7 | 0 | 0 | 0 | 0 | 36
PHARYNGITIS (Infections and infestations) | 2 | 1 | 3 | 1 | 0 | 0 | 0 | 6
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 7 | 9 | 0 | 1 | 0 | 0 | 0 | 16
FALL (Injury, poisoning and procedural complications) | 5 | 0 | 3 | 1 | 0 | 0 | 0 | 7
LIGAMENT SPRAIN (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 2
LIP INJURY (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
BLOOD CHOLESTEROL INCREASED (Investigations) | 6 | 4 | 5 | 1 | 0 | 0 | 0 | 14
BLOOD CREATININE INCREASED (Investigations) | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 3
LIPASE INCREASED (Investigations) | 8 | 2 | 7 | 0 | 0 | 0 | 0 | 15
DECREASED APPETITE (Metabolism and nutrition disorders) | 2 | 2 | 1 | 1 | 0 | 0 | 0 | 6
HYPERCHOLESTEROLAEMIA (Metabolism and nutrition disorders) | 2 | 3 | 7 | 0 | 0 | 0 | 0 | 10
HYPERTRIGLYCERIDAEMIA (Metabolism and nutrition disorders) | 1 | 0 | 1 | 3 | 0 | 0 | 0 | 4
HYPOPHOSPHATAEMIA (Metabolism and nutrition disorders) | 16 | 2 | 5 | 0 | 0 | 0 | 0 | 17
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 17 | 23 | 4 | 0 | 0 | 0 | 0 | 39
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 3
BACK PAIN (Musculoskeletal and connective tissue disorders) | 9 | 7 | 3 | 1 | 0 | 0 | 0 | 19
BONE PAIN (Musculoskeletal and connective tissue disorders) | 4 | 9 | 2 | 0 | 0 | 0 | 0 | 13
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 7 | 4 | 4 | 1 | 0 | 0 | 0 | 14
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 6 | 7 | 0 | 1 | 0 | 0 | 0 | 14
MYALGIA (Musculoskeletal and connective tissue disorders) | 3 | 9 | 3 | 1 | 1 | 0 | 0 | 15
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 8 | 13 | 1 | 1 | 0 | 0 | 0 | 22
ROTATOR CUFF SYNDROME (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 3
AMNESIA (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
HEADACHE (Nervous system disorders) | 9 | 11 | 6 | 1 | 0 | 0 | 0 | 24
ANXIETY (Psychiatric disorders) | 1 | 3 | 0 | 1 | 0 | 0 | 0 | 4
DEPRESSION (Psychiatric disorders) | 3 | 1 | 1 | 1 | 0 | 0 | 0 | 5
MENSTRUATION IRREGULAR (Reproductive system and breast disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 2
COUGH (Respiratory, thoracic and mediastinal disorders) | 7 | 1 | 1 | 1 | 0 | 0 | 0 | 10
DYSPHONIA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 6 | 1 | 1 | 1 | 0 | 0 | 0 | 8
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 3 | 1 | 0 | 0 | 0 | 9
DRY SKIN (Skin and subcutaneous tissue disorders) | 5 | 1 | 0 | 1 | 0 | 0 | 0 | 7
PRURITUS (Skin and subcutaneous tissue disorders) | 4 | 2 | 8 | 1 | 0 | 0 | 0 | 15
RASH (Skin and subcutaneous tissue disorders) | 7 | 1 | 3 | 2 | 0 | 0 | 0 | 13
HYPERTENSION (Vascular disorders) | 16 | 7 | 3 | 1 | 0 | 0 | 0 | 24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigators are NOT employed by the organization sponsoring the study. Other disclosure agreement that restricts the right of the PI to discuss or publish trial results after the trial is completed. The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of pooled data (i.e.,data from all sites) in clinical trial.